CLINICAL TRIAL: NCT02548754
Title: TRanscutaneous Electrical vAgus Nerve sTimulation to Suppress Atrial Fibrillation
Acronym: TREAT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRCH135160; 15MCPRP25790001 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation; Inflammation
Keywords: atrial fibrillation; neuromodulation; inflammation
MeSH Terms: conditions — Atrial Fibrillation; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Patients will receive 1 hour of active low level tragus stimulation daily for 6 months
  Interventions: Device: Parasym device
- Sham (Sham Comparator): Patients will receive 1 hour of sham low level tragus stimulation daily for 6 months
  Interventions: Device: Parasym device

INTERVENTIONS:
Device: Parasym device

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia. In previous experimental studies, the investigators found that low-level vagus nerve (VN) stimulation (LLVNS), at voltages substantially below that which slowed the sinus rate, significantly suppressed AF inducibility and decreased AF duration. The investigators subsequently developed a non-invasive neuromodulatory therapy, in which LLVNS was delivered to the auricular branch of the VN located at the tragus, the anterior protuberance of the outer canine ear (low level tragus stimulation; LLTS). The anti-arrhythmic effects of LLTS were similar to those of LLVNS delivered to the cervical VN trunk. More recently, in a proof-of-concept study in humans, the investigators showed that in patients with drug-refractory AF undergoing AF ablation, LLTS for just one hour significantly shortened the AF duration and decreased inflammatory cytokines.

The overall objective of this proposal is to translate in ambulatory patients with paroxysmal AF the results of previous studies showing acute suppression of AF and inflammation in anesthetized canines as well as humans, in order to examine the long-term therapeutic effects of this approach. The investigators hypothesize that intermittent (1 hour daily) LLTS for 6 months may result in long-term decrease of AF burden and suppression inflammatory cytokines in patients with paroxysmal AF. Patients will be randomized to either active or sham LLTS. LLTS will be delivered through a transcutaneous electrical nerve stimulation (TENS) device for 1 hour daily over a 6-month period. AF burden will be defined as the percent of time spent in AF over a 2-week period, assessed by noninvasive continuous ECG monitoring at baseline and at 6 months. In addition, blood samples will be collected from patients at baseline, and at 3 and 6 months, for cytokine measurement. These investigations will establish the first evidence of the long-term effects of LLTS on AF suppression in patients with paroxysmal AF and may provide the basis for a potential expansion of the therapeutic targets of this treatment modality beyond AF.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients older than 21 year old
2. Paroxysmal AF

Exclusion Criteria:

1. Left ventricular dysfunction (Left ventricular ejection fraction <40%)
2. Significant valvular disorder (i.e., prosthetic valve or hemodynamically relevant valvular diseases)
3. Recent (<6 months) stroke or myocardial infarction
4. Severe heart failure (NYHA IV)
5. Left atrial dilatation (>55mm)
6. Recurrent vaso-vagal syncopal episodes
7. Unilateral or bilateral vagotomy
8. Pregnancy or breast feeding
9. Sick sinus syndrome, 2nd or 3rd degree AV block, bifascicular block or prolonged (PR>300ms) 1st degree AV block.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Stavrakis S, Stoner JA, Humphrey MB, Morris L, Filiberti A, Reynolds JC, Elkholey K, Javed I, Twidale N, Riha P, Varahan S, Scherlag BJ, Jackman WM, Dasari TW, Po SS. TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial. JACC Clin Electrophysiol. 2020 Mar;6(3):282-291. doi: 10.1016/j.jacep.2019.11.008. Epub 2020 Jan 29. PMID 32192678

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Patients will receive 1 hour of active low level tragus stimulation daily for 6 months
  Parasym device
- Sham: Patients will receive 1 hour of sham low level tragus stimulation daily for 6 months
  Parasym device
Period: Overall Study
Arm/Group | Active | Sham
Started | 26 | 27
Completed | 24 | 23
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (15) | 68 (11) | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
AF burden [Median (Inter-Quartile Range); unit: %] | 4.5 [0.2 to 31] | 1 [0 to 15] | 2.5 [0.2 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation Burden
Description: Percent time spent in atrial fibrillation
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Percent time spent in atrial fibrillatio
Arm/Group | Active | Sham
Number analyzed (Participants) | 26 | 27
Percent time spent in atrial fibrillatio | 2 [0 to 11] | 8.5 [0 to 42]

2. Secondary Outcome: Markers of Inflammation
Description: Serum levels of tumor necrosis factor-alpha
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Active | Sham
Number analyzed (Participants) | 26 | 27
pg/ml | 5.5 [3.9 to 8.3] | 5.4 [4.4 to 8.3]

3. Secondary Outcome: Markers of Inflammation
Description: Serum levels of inteleukin 6
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Active | Sham
Number analyzed (Participants) | 26 | 27
pg/ml | 1.5 [0.7 to 3.2] | 2.3 [1 to 4.4]

ADVERSE EVENTS:
Time Frame: 6 months
Description: No device related adverse events reported
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 1/26 | 2/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02548754/Prot_SAP_001.pdf